CLINICAL TRIAL: NCT04239833
Title: A Phase III, Double-blind, Randomised Study of SH-1028 Tablets Versus Gefiitinib as First Line Treatment in Patients With Epidermal Growth Factor Receptor Mutation Positive, Locally Advanced or Metastatic Non Small Cell Lung Cancer
Brief Title: A Study of SH-1028 Tablets Versus Gefitinib in Patients With Locally Advanced or Metastatic Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nanjing Sanhome Pharmaceutical, Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SHC013-III-01
Record Dates: First submitted 2020-01-02; First posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2019-12

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — SH-1028; Gefitinib

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to SH-1028 tablets arm or Gefitinib arm based on the mutation condition of EGFR (L858R or 19Del) and brain metastases (yes or no). The rate of SH-1028 tablets arm to Gefitinib arm is 2:1.
Who Masked: Participant, Care Provider, Investigator
Masking Description: All trial personnel and participants were masked to treatment allocation, until unblinding due to progression disease or other Criteria of termination.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SH-1028 tablets+Placebo Gefitinib (Experimental): SH-1028 tablets (200 mg orally, once daily) plus placebo Gefitinib (250 mg orally, once daily), in accordance with the randomization schedule.
  Interventions:
  Drug: SH-1028 tablets 200 mg Drug: Placebo Gefitinib 250 mg
  Interventions: Drug: SH-1028 tablets; Drug: Placebo Gefitinib
- Gefitinib+Placebo SH-1028 tablets (Active Comparator): Gefitinib (250 mg orally, once daily) plus placebo SH-1028 tablets (200mg orally, once daily), in accordance with the randomisation schedule.
  Following objective disease progression according to RECIST 1.1, as per investigator assessment, patients who were randomized to Standard of Care arm may have the option to receive open-label SH-1028 tablets (crossover to active SH-1028 tablets).
  Interventions:
  Drug: Gefitinib 250 mg Drug: Placebo SH-1028 tablets 200mg
  Interventions: Drug: Placebo SH-1028 tablets; Drug: Gefitinib

INTERVENTIONS:
Drug: SH-1028 tablets — The initial dose of SH-1028 tablets is 200 mg once daily . A cycle of treatment is defined as 21 days of once daily treatment.
  Number of Cycles: as long as patients are continuing to show clinical benefit, as judged by the Investigator, and in the absence of discontinuation criteria.
  Arms: SH-1028 tablets+Placebo Gefitinib
Drug: Placebo SH-1028 tablets — The initial dose of Placebo SH-1028 tablets is 200 mg once daily . A cycle of treatment is defined as 21 days of once daily treatment.
  Number of Cycles: as long as patients are continuing to show clinical benefit, as judged by the Investigator, and in the absence of discontinuation criteria.
  Arms: Gefitinib+Placebo SH-1028 tablets
Drug: Gefitinib — The initial dose of Gefitinib is 250 mg once daily . A cycle of treatment is defined as 21 days of once daily treatment.
  Following objective disease progression according to RECIST 1.1, as per investigator assessment, patients who were randomized to Standard of Care arm may have the option to receive open-label SH-1028 tablets (crossover to active SH-1028 tablets).
  Arms: Gefitinib+Placebo SH-1028 tablets
Drug: Placebo Gefitinib — The initial dose of Gefitinib is 250 mg once daily . A cycle of treatment is defined as 21 days of once daily treatment.
  Arms: SH-1028 tablets+Placebo Gefitinib

SUMMARY:
To assess the efficacy and safety of SH-1028 tablets versus Gefitinib, a standard of care epidermal growth factor receptor tyrosine kinase inhibitor, in patients with locally advanced or Metastatic Non Small Cell Lung Cancer

DETAILED DESCRIPTION:
This is a Phase III, multi-center,double-blind, randomised study assessing the efficacy and safety of SH-1028 tablets (200 mg orally, once daily) versus a standard of care (SoC) Epidermal Growth Factor Receptor (EGFR) Tyrosine Kinase Inhibitor (TKI) ( gefitinib, 250 mg orally, once daily) in patients with locally advanced or metastatic Non-small Cell Lung Cancer (NSCLC) that is known to be EGFR sensitising mutation (EGFRm) positive, treatment-naive and eligible for first-line treatment with an EGFR-TKI.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female, aged at least 18 years.
* 2. Pathologically or cytologically confirmed locally advanced or metastatic NSCLC (e.g. this may occur systemic recurrence after prior surgery for early stage disease or patients may be newly diagnosed with stage IIIB/IV disease). Patients must be treatment-naïve for locally advanced or metastatic NSCLC. Prior adjuvant and neo-adjuvant therapy is permitted (chemotherapy, radiotherapy, investigational agents) provided all other entry criteria are satisfied.
* 3. The tumour harbours one of the 2 common EGFR mutations known to be associated with EGFR-TKI sensitivity (Ex19del, L858R), either or in combination with other EGFR mutations assessed by central testing using tumour tissue sample or cytology sample.
* 4. A ECOG performance status equal to 0-1 with a minimum life expectancy of 12 weeks.
* 5. At least 1 lesion that has not previously been irradiated, that has not been chosen for biopsy during the study screening period, and that can be accurately measured at Baseline as ≥ 10 mm in the longest diameter (except lymph nodes, which must have short axis ≥ 15mm) with computerized tomography (CT) or magnetic resonance imaging (MRI), whichever is suitable for accurately repeated measurements.
* 6. Adequate bone marrow reserve or organ function, as demonstrated by the following laboratory values:

  1. Absolute neutrophil count (ANC）≥1.5×10^9 / L
  2. Platelet count ≥100×10^9 / L
  3. Hemoglobin ≥90 g/L
  4. Alanine aminotransferase (ALT) ≤ 2.5 × upper limit of normal (ULN) if no demonstrable liver metastases or ≤ 5 × ULN in the presence of liver metastases.
  5. Aspartate aminotransferase (AST) ≤ 2.5 × ULN if no demonstrable liver metastases or ≤ 5 × ULN in the presence of liver metastases.
  6. Total bilirubin (TBL) ≤ 1.5 × ULN if no liver metastases or ≤ 3 × ULN in the presence of documented Gilbert's Syndrome (unconjugated hyperbilirubinemia) or liver metastases.
  7. Creatinine ≤ 1.5 × ULN concurrent with creatinine clearance ≥ 50 mL/min (measured or calculated by the Cockcroft-Gault equation); confirmation of creatinine clearance is only required when creatinine is ≤ 1.5 × ULN.
* 7. Females of child-bearing potential should be using adequate contraceptive measures throughout the study, should not be breast feeding during the study and until 6 months after completion of study, and must have a negative pregnancy test prior to start of dosing.
* 8. Male patients should be willing to use barrier contraception during the study and until 6 months after completion of study (i.e., condoms).
* 9. Do not participate in other clinical trial (enroll and take medicine) in 1 month prior to start of dosing.
* 10.Patients must sign and date written informed consent prior to admission to the study.

Exclusion Criteria:

* 1. Treatment with any of the following, including any EGFR-TKI, systemic chemotherapy (except for relapsed patients at last 6 months after received post-surgery adjuvant chemotherapy)，immunotherapy, targeted therapy and anti-tumor traditional Chinese medicine therapy.
* 2. Major surgery (excluding placement of vascular access) within 4 weeks of the first dose of study drug.
* 3. Radiotherapy with a limited field of radiation for palliation within 1 week of the first dose of study drug, with the exception of patients receiving radiation to > 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of study drug.
* 4. The patient is currently using (or cannot discontinue at least 1 week before the first dose of study drug) a drug or herbal supplement known as a potent inhibitor or inducer of CYP3A4.
* 5. Treatment with large doses of glucocorticoids (eg, >10 mg/day dexamethasone ) or other immunosuppressive agents within 2 weeks.
* 6. Any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE), Grade 1, at the time of starting study treatment with the exception of alopecia and Grade 2, prior platinum-therapy related neuropathy.
* 7. Spinal cord compression, meningeal metastases or brain metastases unless asymptomatic, s table, and not requiring steroids for at least 4 weeks prior to start of study treatment.
* 8. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension or active bleeding diatheses, or which in the Investigator's opinion makes it undesirable for the patient to participate in the trial.
* 9. Active infection (e.g., hepatitis B, hepatitis C or human immunodeficiency virus [HIV]). (HBsAg is positive but HBV-DNA < ULN, and HCVAb is positive but HCV-RNA<ULN can be accepted.）
* 10. Any of the following cardiac criteria:

  1. Mean resting corrected QT interval (QTcF) > 470 msec obtained from 3 electrocardiograms (ECGs), using the Screening clinic ECG machine and Fridericia's formula for QT interval correction.
  2. Any clinically important abnormalities in rhythm, conduction, or morphology of the resting ECG (e.g., complete left bundle branch block, third-degree heart block, second-degree heart block, PR interval >250 msec).
  3. Any factors that increase the risk of QTc prolongation or risk of arrhythmic events, such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome, or unexplained sudden death under 40 years of age in first degree relatives or any concomitant medication known to prolong the QT interval.
  4. Left ventricular ejection fraction (LVEF) ≤ 40%.
* 11. Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease.
* 12. History of any other malignant tumor within five years (except clinically cured cervical carcinoma in situ, basal cells or squamous epithelial skin cancer).
* 13. Any seriously abnormal gastrointestinal function would affect uptake, transport and absorption of the drug, such as inability to swallow the study medication, refractory nausea and vomiting, previous significant bowel resection, Recurrent diarrhea, atrophic gastritis (age < 60 years), unhealed serious gastric diseases, Crohn's disease or ulcerative colitis.
* 14. History of hypersensitivity to any active or inactive ingredient of SH-1028 or drug with a similar chemical structure or class to SH-1028.
* 15. Any severe and uncontrolled ocular disease that may, in the Investigator's opinion, present a specific risk to the patient's safety.
* 16. Lactating Women.
* 17. Any disease or condition that, in the opinion of the Investigator, would compromise the safety of the patient or interfere with study assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2020-01-31 (Estimated); Primary Completion 2022-01-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Median Progression Free Survival (PFS) | At baseline and every 6 weeks relative to randomisation until progression，up to 24 months.
  Progression-free survival was defined as the time from randomization until the date of objective disease progression regardless of whether the participant withdrew from randomized therapy and was used to assess the efficacy of SH-1028 tablets compared with Gefitinib (SoC EGFR-TKI therapy) as measured by PFS. The primary endpoint of PFS was based on Investigator assessment.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | At baseline and every 6 weeks relative to randomisation until progression，up to 24 months.
  ORR was defined as the number (%) of participants with measurable disease with at least 1 visit response of Complete response (CR) or Partial response (PR) and it was used to further assess the efficacy of SH-1028 tablets compared with Gefitinib (SoC EGFR-TKI therapy). ORR was based on Investigator assessment.
Duration of Response (DoR) | At baseline and every 6 weeks relative to randomisation until progression，up to 24 months.
  Duration of response was defined as the time from the date of first documented response until the date of documented progression or death in the absence of disease progression and was used to further assess the efficacy of SH-1028 tablets compared with Gefitinib (SoC EGFR-TKI therapy).
Disease Control Rate (DCR) | At baseline and every 6 weeks relative to randomisation until progression，up to 24 months.
  The DCR was defined as the percentage of participants who had a best overall response (BOR) of Complete response (CR), Partial response (PR) or Stable disease (SD) ≥6 weeks prior to any Progressive disease (PD) event and was used to further assess the efficacy of SH-1028 tablets compared with Gefitinib (SoC EGFR-TKI therapy).
Depth of Response（DepOR） | At baseline and every 6 weeks relative to randomisation until progression，up to 24 months.
  The Depth of response was defined as the relative change in the sum of the longest diameters of Response Evaluation Criteria in Solid Tumors (RECIST) Target lesions (TLs) at the nadir, in the absence of new lesions (NLs) or progression of Non-target lesions (NTLs), compared to baseline and was used to further assess the efficacy of SH-1028 tablets compared with Gefitinib (SoC EGFR-TKI therapy).
Overall Survival (OS) | From first dose to end of study or date of death from any cause, whichever comes first, assessed every 6 weeks (approximately 30 months)
  Overall survival was defined as the time from the date of randomisation until death from any cause and was used to further assess the efficacy of SH-1028 tablets compared with Gefitinib (SoC EGFR-TKI therapy).
Change From Baseline in European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life (QLQ) Questionnaires Lung Cancer 13 (QLQ-LC13) | At baseline and every 6 weeks relative to randomisation until progression，up to 24 months.
  The EORTC QLQ-LC13 was a lung-cancer-specific module comprising 13 questions to assess lung cancer symptoms (cough, haemoptysis, dyspnoea, and site-specific pain); treatment related side-effects (sore mouth, dysphagia, peripheral neuropathy, and alopecia); and pain medication. An outcome variable consisting of a score from 0 to 100 was derived for each of the symptom scales/symptom items. Higher scores on the global health status/QoL and functioning scales indicated better health status/QoL and function. Higher scores on the symptoms scales indicated greater symptom burden. The analysis was performed using a Mixed-effects model for repeated measures analysis on the change from baseline in PRO symptom score at each visit, including participants, treatment, visit and treatment by visit interaction as explanatory variables, the baseline PRO score as a covariate along with the baseline PRO score by visit interaction, using an unstructured covariance structure.
Change From Baseline in European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 Items (EORTC QLQ-C30) | At baseline and every 6 weeks relative to randomisation until progression，up to 24 months.
  The EORTC QLQ-C30 cancer-specific questionnaire consisted of 30 questions, combined to produce 5 functional scales, 3 symptom scales, 6 individual items, and a global measure of health status/QoL. An outcome variable consisting of a score from 0 to 100 was derived for each of the symptom scales/symptom items, the functional scales, and the global health status/QoL scale in the EORTC QLQ-C30. Higher scores on the global health status and functioning scales indicated better health status/function. Higher scores on the symptoms scales indicated greater symptom burden. The analysis was performed using a Mixed-effects model for repeated measures analysis on the change from baseline in PRO symptom score at each visit, including participants, treatment, visit and treatment by visit interaction as explanatory variables, the baseline PRO score as a covariate along with the baseline PRO score by visit interaction, using an unstructured covariance structure.
Number of adverse events (AEs) | From first dose to 28 days after SH-1028 tablets discontinuation.
  Number of adverse events (AEs) assessed by CTCAE 5.0 was one of main outcome measures to compare the safety of SH-1028 Tablets and Gefitinib.
Incidence rate of serious adverse events (SAEs) | From first dose to 28 days after SH-1028 tablets discontinuation.
  Incidence rate of serious adverse events (SAEs) was one of main outcome measures to compare the safety of SH-1028 Tablets and Gefitinib.

CONTACTS AND LOCATIONS:
Overall Officials: Zhou Caicun, Professor, Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No